CLINICAL TRIAL: NCT00835978
Title: Randomized, Double-blind Phase 2 Study Of Axitinib (Ag-013736) With Or Without Dose Titration In Patients With Metastatic Renal Cell Carcinoma
Brief Title: Axitinib (AG-013736) With Or Without Dose Titration (Increase) In Patients With Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A4061046; 2008-007786-23 (EudraCT Number)
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Carcinoma, Renal Cell
Keywords: axitinib or AG-013736 dose titration (increase) renal cell carcinoma; kidney cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Axitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Other): Randomized arm
  Interventions: Drug: axitinib
- B (Other): Randomized arm
  Interventions: Drug: axitinib
- C (Other): Non-randomized arm
  Interventions: Drug: axitinib

INTERVENTIONS:
Drug: axitinib — axitinib 5mg BID (open-label) + axitinib dose titration (blinded)
  Arms: A
Drug: axitinib — axitinib 5mg BID (open-label) + placebo dose titration (blinded)
  Arms: B
Drug: axitinib — axitinib 5mg BID (open-label)
  Arms: C

SUMMARY:
Axitinib dose titration (giving a higher dose of the drug above its standard starting dose) among certain patients may improve the response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* metastatic renal cell carcinoma (kidney cancer) with clear cell component
* no prior systemic therapy (including no prior adjuvant or neoadjuvant)
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Blood Pressure < or = 140/90mmHg

Exclusion Criteria:

* brain/CNS metastasis
* using more than 2 blood pressure medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2009-08; Primary Completion 2012-10 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (64):
- United States (31):
  - East Bay Medical Oncology/Hematology Medical Associates Inc., Antioch, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Bay Area Cancer Research Group, LLC, Pleasant Hill, California
  - Diablo Valley Oncology and Hematology Medical Group Inc, Pleasant Hill, California
  - East Bay Medical Oncology/Hematology Medical Associates Inc, Pleasant Hill, California
  - East Bay Medical Oncology/Hematology Medical Associates Inc, San Leandro, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Investigational Drug Services, IUHSCC, Indianapolis, Indiana
  - IU Health University Hospital, Indianapolis, Indiana
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Institute, Las Vegas, Nevada
  - The University Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, James Cancer Hospital, Columbus, Ohio
  - JamesCare in Kenny, Columbus, Ohio
  - West Chester Hospital Medical Building, West Chester, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Texas Oncology, Sammons Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington
- Czechia (4):
  - Masarykuv onkologicky ustav, Brno, CZE
  - Fakultni nemocnice Olomouc Onkologicka klinika, Olomouc
  - Fakultni nemocnice Na Bulovce, Prague
  - Krajska zdravotni, a.s. - Masarykova nemocnice V Usti nad Labem, o.z., Ústí nad Labem
- Germany (5):
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Klinikum der J. W. Goethe-Universitaet, Medizinische Klinik II, Frankfurt
  - Medizinische Hochschule Hannover, Abt. Haematologie, Haemostaseologie & Onkologie, Hanover
  - Eberhardt-Karls-Universitaet Tuebingen, Klinik fuer Urologie, Tübingen
  - Klinikum Weiden Klinik fuer Urologie, Andrologie und Kinderurologie, Weiden
- Japan (15):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Kinki University Hospital, Sayama, Osaka
  - Hamamatsu University School of Medicine, University Hospital, Hamamatsu, Shizuoka
  - National Cancer Center, Chuo-ku, Tokyo
  - Japanese Foundation For Cancer Research Cancer Institute Hospital, Koto-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Akita University Hospital, Akita
  - Chiba Cancer Center, Chiba
  - Kyushu University Hospital, Fukuoka
  - Nagasaki University Hospital, Nagasaki
  - Tokushima University Hospital, Tokushima
  - Yamagata University Hospital, Yamagata
- Russia (6):
  - Medical Radiology Research Center of the Minzdravsotsrazvitiya of Russia, Obninsk, Kaluga Oblast
  - State Healthcare Institution "Leningrad Regional Oncology Dispensary", Poselok Kuzmolovskiy, Vsevolozhskiy Region, Leningradskaya Oblast
  - FSBSI "N.N. Blokhin Russian Cancer Research Center", Moscow
  - FSBI"Russian Scientific Center of Roengenoradiology" of the MH of RF, Moscow
  - Saint-Petersburg's State Healthcare Institution 'City Clinical Oncology Dispensary', Saint Petersburg
  - GBUZ "Samara Regional Clinical Oncology Dispensary", Samara
- Spain (3):
  - Hospital de La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid

REFERENCES:
- [Derived] Tomita Y, Uemura H, Oya M, Shinohara N, Habuchi T, Fujii Y, Kamei Y, Umeyama Y, Bair AH, Rini BI. Patients with metastatic renal cell carcinoma who benefit from axitinib dose titration: analysis from a randomised, double-blind phase II study. BMC Cancer. 2019 Jan 7;19(1):17. doi: 10.1186/s12885-018-5224-6. PMID 30616534
- [Derived] de Velasco G, McKay RR, Lin X, Moreira RB, Simantov R, Choueiri TK. Comprehensive Analysis of Survival Outcomes in Non-Clear Cell Renal Cell Carcinoma Patients Treated in Clinical Trials. Clin Genitourin Cancer. 2017 Dec;15(6):652-660.e1. doi: 10.1016/j.clgc.2017.03.004. Epub 2017 Mar 21. PMID 28410911
- [Derived] Grunwald V, Lin X, Kalanovic D, Simantov R. Early Tumour Shrinkage: A Tool for the Detection of Early Clinical Activity in Metastatic Renal Cell Carcinoma. Eur Urol. 2016 Dec;70(6):1006-1015. doi: 10.1016/j.eururo.2016.05.010. Epub 2016 May 26. PMID 27238653
- [Derived] Rini BI, Melichar B, Ueda T, Grunwald V, Fishman MN, Arranz JA, Bair AH, Pithavala YK, Andrews GI, Pavlov D, Kim S, Jonasch E. Axitinib with or without dose titration for first-line metastatic renal-cell carcinoma: a randomised double-blind phase 2 trial. Lancet Oncol. 2013 Nov;14(12):1233-42. doi: 10.1016/S1470-2045(13)70464-9. Epub 2013 Oct 18. PMID 24140184
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061046&StudyName=Axitinib%20%28AG-013736%29%20With%20Or%20Without%20Dose%20Titration%20%28Increase%29%20In%20Patients%20With%20Kidney%20Cancer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 49 centers in Czech Republic, Germany, Japan, Russian Federation, Spain, and the United States (US).
Pre-assignment Details: Participants were enrolled in a 4-week lead-in period, during which they received axitinib 5 milligram (mg) twice a day (BID). After the lead-in period, participants meeting randomization criteria were then randomized to one of the two treatment arms. Participants, not meeting criteria, continued study without dose titration (non-randomized arm).
Groups:
- Active Titration Arm: Participants initially received axitinib 5 mg twice a day (BID) + axitinib (blinded therapy) 2 mg BID. After at least 2 consecutive weeks, participants satisfying the dose titration criteria had their dose level increased by one additional dose level, to axitinib 5 mg BID + axitinib (blinded therapy) 5 mg BID, unless otherwise contraindicated per the investigator's clinical judgment. The maximum total daily dose was 10 mg BID (axitinib 5mg BID + axitinib [blinded therapy] 5 mg BID).
- Placebo Titration Arm: Participants initially received axitinib 5mg BID + placebo (blinded therapy) 2 mg BID. After at least 2 consecutive weeks, participants satisfying the dose titration criteria had their dose level increased by one additional dose level, to axitinib 5 mg BID + placebo (blinded therapy) 5 mg BID, unless otherwise contraindicated per the investigator's clinical judgment. The maximum total daily dose was 10 mg BID (axitinib 5mg BID + placebo [blinded therapy] 5 mg BID).
- Non-randomized Arm: Participants not eligible for randomization were assigned to receive axitinib 5 mg BID or a reduced dose per the dose modification guideline. Dose titration was not permitted in this treatment arm.
- Discontinued Prior to Randomization: Participants who discontinued before they were randomized to any of the treatment or non-randomized arms.
Period: Overall Study
Arm/Group | Active Titration Arm | Placebo Titration Arm | Non-randomized Arm | Discontinued Prior to Randomization
Started | 56 | 56 | 91 | 10
Treated | 56 | 56 | 91 | 10
Completed | 0 (Study Completion: 29 Feb 2016. Treatment discontinued due to objective progression/relapse & death) | 0 (Study Completion: 29 Feb 2016. Treatment discontinued due to objective progression/relapse & death) | 0 (Study Completion: 29 Feb 2016. Treatment discontinued due to objective progression/relapse & death) | 0 (Study Completion: 29 Feb 2016. Treatment discontinued due to objective progression/relapse & death)
Not Completed | 56 | 56 | 91 | 10
Not completed — Death | 33 | 40 | 49 | 4
Not completed — Lost to Follow-up | 3 | 4 | 2 | 1
Not completed — Other | 5 | 1 | 8 | 0
Not completed — Objective progression or relapse | 2 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 5
Not completed — Study terminated by sponsor | 12 | 8 | 30 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis (SA) population consists of all participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Titration Arm | Placebo Titration Arm | Non-randomized Arm | Discontinued Prior to Randomization | Total
Number analyzed (Participants) | 56 | 56 | 91 | 10 | 213
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.7 (10.2) | 59.6 (10.5) | 62.9 (8.9) | 62.9 (7.5) | 61.2 (9.7)
Age, Customized [Number; unit: Participants]
  < 65 Years | 38 | 38 | 54 | 6 | 136
  >= 65 Years | 18 | 18 | 37 | 4 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 11 | 36 | 4 | 70
  Male | 37 | 45 | 55 | 6 | 143

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) - Percentage of Participants With Objective Response
Description: ORR was defined as the proportion of participants with objective response based assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.0). CR was defined as complete disappearance of all target lesions and non-target disease. No new lesions. PR was defined as >=30% decrease on study under baseline of the sum of longest diameters of all target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Baseline up to disease progression, death, or withdrawal; performed at baseline and repeated every 8 weeks for 24 weeks, then every 12 weeks.
Population: The Full Analysis (FA) population included all randomized participants who received study drug or different drug to which they were randomized. The Safety Analysis (SA) population included all non-randomized patients who received at least 1 dose of study medication with treatment assignments designated according to actual study treatment received.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- All Participants: All enrolled participants (randomized and non-randomized)
Arm/Group | Active Titration Arm | Placebo Titration Arm | Non-randomized Arm | All Participants
Number analyzed (Participants) | 56 | 56 | 91 | 213
Percentage of Participants | 53.6 [39.7 to 67.0] | 33.9 [21.8 to 47.8] | 59.3 [48.5 to 69.5] | 48.4 [41.5 to 55.3]
Statistical Analysis 1: Comparison: Active Titration Arm vs Placebo Titration Arm; ORR for the 2 treatment arms was compared with the Cochran-Mantel-Haenszel test stratified by ECOG performance status. The relative risk ratio estimator was used to contrast the treatment effects on the endpoint. Both a point estimate and a 2-sided 95% CI were calculated using a normal approximation; Test type: Superiority or Other; p = 0.0189, Cochran-Mantel-Haenszel — A priori defined threshold for statistical significance was: alpha=0.10 (one-sided); Risk Ratio (RR) = 1.578, 95% CI 2-sided [1.017 to 2.448]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: The time from first dose administration to first documentation of objective tumor progression or to death due to any cause. PFS in each arm was assessed using the Kaplan-Meier method and estimates of the PFS curves from the Kaplan-Meier method were presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Active Titration Arm | Placebo Titration Arm | Non-randomized Arm | All Participants
Number analyzed (Participants) | 56 | 56 | 91 | 213
Months | 14.5 [9.2 to 24.5] | 15.7 [8.3 to 19.4] | 16.6 [11.2 to 22.5] | 14.6 [11.5 to 17.5]
Statistical Analysis 1: Comparison: Active Titration Arm vs Placebo Titration Arm; Test type: Superiority or Other; p = 0.2444, Log Rank; Hazard Ratio (HR) = 0.849, 95% CI 2-sided [0.535 to 1.348]

3. Secondary Outcome: Duration of Response (DR)
Description: DR was defined as the time from the first documentation of objective tumor response (complete response - CR or Partial response - PR) to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first. The median values were estimated based on Kaplan-Meier method. 95% confidence interval was based on the Brookmeyer and Crowley method.
Time Frame: as for outcome 1
Population: Subset of Full Analysis (FA) and Safety Analysis (SA) patients who achieved confirmed complete or partial response. FA included all randomized patients and was based on randomized treatment assignment regardless of whether or not study drug was administered. SA included all non randomized patients who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Active Titration Arm: Participants initially received axitinib 5 mg twice a day (BID) + axitinib(blinded therapy) 2 mg BID. After at least 2 consecutive weeks, participants satisfying the dose titration criteria had their dose level increased by one additional dose level, to axitinib 5 mg BID + axitinib (blinded therapy) 5 mg BID, unless otherwise contraindicated per the investigator's clinical judgment. The maximum total daily dose was 10 mg BID (axitinib 5mg BID + axitinib [blinded therapy] 5 mg BID).
Arm/Group | Active Titration Arm | Placebo Titration Arm | Non-randomized Arm
Number analyzed (Participants) | 30 | 19 | 54
Months | NA [10.8 to NA] — The median duration of tumor response among responders was not reached in the active treatment group. | 21.2 [11.1 to 25.8] | 23.3 [15.7 to 28.6]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of the first dose of the study medication to date of death due to any cause. For participants who did not die, their survival times were to be censored at the last date they were known to be alive.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Active Titration Arm (FA Population): Participants initially received axitinib 5 mg twice a day (BID) + axitinib (blinded therapy) 2 mg BID. After at least 2 consecutive weeks, participants satisfying the dose titration criteria had their dose level increased by one additional dose level, to axitinib 5 mg BID + axitinib (blinded therapy) 5 mg BID, unless otherwise contraindicated per the investigator's clinical judgment. The maximum total daily dose was 10 mg BID (axitinib 5mg BID + axitinib [blinded therapy] 5 mg BID).
- Placebo Titration Arm (FA Population): Participants initially received axitinib 5mg BID + placebo (blinded therapy) 2 mg BID. After at least 2 consecutive weeks, participants satisfying the dose titration criteria had their dose level increased by one additional dose level, to axitinib 5 mg BID + placebo (blinded therapy) 5 mg BID, unless otherwise contraindicated per the investigator's clinical judgment. The maximum total daily dose was 10 mg BID (axitinib 5mg BID + placebo [blinded therapy] 5 mg BID).
- Non-randomized Arm (SA Population): Participants not eligible for randomization were assigned to receive axitinib 5 mg BID or a reduced dose per the dose modification guideline. Dose titration was not permitted in this treatment arm.
Arm/Group | Active Titration Arm (FA Population) | Placebo Titration Arm (FA Population) | Non-randomized Arm (SA Population)
Number analyzed (Participants) | 56 | 56 | 91
Months | 42.7 [24.7 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times | 30.4 [23.7 to 45.0] | 41.6 [33.0 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Axitinib
Description: Cmax for steady-state axitinib was evaluated on Cycle 2 Day 15. Results were normalized to axitinib 7 mg dose for active titration arm and axitinib 5 mg dose for placebo titration arm. Results were normalized to axitinib 7 mg dose for active titration arm and axitinib 5 mg dose for placebo titration arm.
Time Frame: Cycle 2 Day 15 (C2D15): pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose
Population: The pharmacokinetic (PK) population included all participants who were treated and had at least 1 concentration on 1 PK assessment day. The PK parameter analysis data set included all participants treated who had at least 1 estimated PK parameter of primary interest.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Active Titration Arm | Placebo Titration Arm
Number analyzed (Participants) | 16 | 20
ng/mL | 31.74 [21.63 to 46.58] | 23.05 [16.36 to 32.49]

6. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Axitinib,
Description: Tmax for steady-state axitinib was evaluated on Cycle 2 Day 15.
Time Frame: C2D15: pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose
Population: as for outcome 5
Measure: Median (Full Range); unit: hrs
Arm/Group | Active Titration Arm | Placebo Titration Arm
Number analyzed (Participants) | 16 | 20
hrs | 2.04 [1.00 to 6.00] | 2.00 [0.00 to 6.00]

7. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Axitinib
Description: Area under the plasma concentration time-curve from zero to the last measurable concentration (AUClast). AUClast for steady-state axitinib was evaluated on Cycle 2 Day 15. Results were normalized to axitinib 7 mg dose for active titration arm and axitinib 5 mg dose for placebo titration arm.
Time Frame: C2D15: pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: ng.hr/mL
Arm/Group | Active Titration Arm | Placebo Titration Arm
Number analyzed (Participants) | 16 | 20
ng.hr/mL | 105.33 [70.16 to 158.14] | 78.44 [54.53 to 112.82]

8. Secondary Outcome: Area Under the Curve From Time Zero to 24 Hours[AUC(0-24)] for Axitinib
Description: Area under the plasma concentration time-curve from zero 24 hours[AUC(0-24). AUC(0-24) for steady-state axitinib was evaluated on Cycle 2 Day 15. Results were normalized to axitinib 7 mg dose for active titration arm and axitinib 5 mg dose for placebo titration arm.
Time Frame: C2D15: pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: ng.hr/mL
Arm/Group | Active Titration Arm | Placebo Titration Arm
Number analyzed (Participants) | 16 | 20
ng.hr/mL | 258.68 [150.47 to 444.72] | 161.38 [102.09 to 255.12]

9. Secondary Outcome: Plasma Decay Half-Life (t1/2) for Axitinib
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Plasma decay half life for steady-state axitinib was evaluated on Cycle 2 Day 15.
Time Frame: C2D15: pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr
Groups:
- Placebo Titration Arm: Participants initially received axitinib 5mg BID + placebo (blinded therapy) 2 mg BID. After at least 2 consecutive weeks, participants satisfying the dose titration criteria had their dose level increased by one additional dose level, to axitinib 5 mg BID + placebo (blinded therapy) 5 mg BID, unless otherwise contraindicated per the investigator's clinical judgment. The maximum total daily dose was 10 mg BID (axitinib 5mg BID + placebo[blinded therapy] 5 mg BID).
Arm/Group | Active Titration Arm | Placebo Titration Arm
Number analyzed (Participants) | 16 | 20
hr | 2.48 (1.902) | 2.81 (1.685)

10. Secondary Outcome: Apparent Oral Clearance (CL/F) of Axitinib
Description: Clearance (CL) of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed (F). Clearance is defined as the volume of blood from which drug can be completely removed per unit of time. CL/F for steady-state axitinib was evaluated on Cycle 2 Day 15.
Time Frame: C2D15: pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: L/hr
Arm/Group | Active Titration Arm | Placebo Titration Arm
Number analyzed (Participants) | 16 | 20
L/hr | 54.15 [31.49 to 93.12] | 61.93 [39.17 to 97.91]

11. Secondary Outcome: Apparent Volume of Distribution During the Elimination Phase (Vz/F) for Axitinib
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Vz/F is influenced by the fraction absorbed. Vz/F for steady-state axitinb was evaluated on Cycle 2 Day 15.
Time Frame: C2D15: pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: L
Arm/Group | Active Titration Arm | Placebo Titration Arm
Number analyzed (Participants) | 16 | 20
L | 158.18 [98.38 to 254.34] | 216.62 [145.00 to 323.60]

12. Secondary Outcome: Change From Baseline in Systolic Blood Pressure
Description: Value at respective visit minus value at baseline
Time Frame: At screening (D-14 to D-1); lead-in period: Cycle 1 - Day 1 and Day 15; Cycle 2 - Day 1 and Day 15; Cycle 3 & subsequent cycles Day 1; end of study and follow-up 28 days after last dose.
Population: The SA population consists of all participatns who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Active Titration Arm | Placebo Titration Arm | Non-randomized Arm
Number analyzed (Participants) | 56 | 56 | 91
mmHg
  Cycle 1 Day 1 (n=52,51,73) | -4.3 (11.1) | -2.9 (9.2) | -1.8 (14.2)
  Cycle 1 Day 15 (n=56,56,91) | 3.8 (12.2) | 4.1 (12.5) | 11.5 (18.0)
  Cycle 2 Day 1 (n=56,56,91) | 1.9 (12.4) | 0.9 (13.6) | 9.9 (18.7)
  Cycle 2 Day 15 (n=55,55,86) | 3.6 (13.8) | 2.7 (16.6) | 5.9 (20.3)
  Cycle 3 Day 1 (n=48,49,84) | 3.5 (15.1) | 8.4 (15.4) | 5.2 (20.2)
  Cycle 4 Day 1 (n=45,48,79) | 4.3 (12.7) | 3.5 (13.0) | 5.5 (18.2)
  End of treatment (n=35,44,51) | 2.4 (17.0) | 1.7 (14.0) | -2.8 (19.0)
  Follow-up (n=16,25,36) | -3.6 (16.9) | -0.4 (16.3) | -0.6 (16.7)

13. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure
Description: Value at respective visit minus value at baseline.
Time Frame: as for outcome 12
Population: The SA population consists of all participatns who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Active Titration Arm | Placebo Titration Arm | Non-randomized Arm
Number analyzed (Participants) | 56 | 56 | 91
mmHg
  Cycle 1 Day 1 (n=52,51,73) | -1.6 (8.2) | -2.6 (7.4) | 0.5 (8.4)
  Cycle 1 Day 15 (n=56,56,91) | 4.8 (8.5) | 3.0 (7.7) | 11.5 (10.0)
  Cycle 2 Day 1 (n=56,56,91) | 4.2 (9.0) | 3.5 (8.0) | 10.5 (10.5)
  Cycle 2 Day 15 (n=55,55,86) | 5.5 (10.5) | 4.4 (10.7) | 9.7 (11.3)
  Cycle 3 Day 1 (n=48,49,84) | 6.6 (8.3) | 5.9 (9.3) | 9.1 (13.6)
  Cycle 4 Day 1 (n=45,48,79) | 7.4 (8.2) | 4.6 (8.5) | 8.7 (11.8)
  End of treatment (n=35,44,51) | 0.6 (10.8) | 3.5 (6.3) | 3.0 (10.5)
  Follow-up (n=16,25,36) | -4.5 (10.1) | -1.3 (8.5) | 1.8 (9.0)

14. Secondary Outcome: Comparison of Circulating Endothelial Cells (CECs) in Blood: Cluster of Differentiation (CD)146+/CD105+ at Baseline
Description: CECs are noninvasive marker of vascular damage, remodeling, and dysfunction. Samples were collected and following proteins were analyzed: CD146+/CD105+ CECs, CD146+/CD105+ mean fluorescence intensity (MFI) platelet derived growth factor receptor (PDGFR)-beta, CD146+/CD105+ MFI phospho-PDGFR (pPDGFR)-beta, CD146+/CD105+ phospho-Vascular endothelial growth factor receptor (pVEGFR), CD146+/CD105+ MFI VEGFR. The ratio of plasma levels of the biomarkers at the selected time point vs baseline is reported.
Time Frame: At baseline - Beginning of the lead-in period (Cycle 1 Day 1)
Population: The Biomarker Analysis Set included participants receiving at least one dose of treatment, with a Cycle 1 Day 1 biomarker result for at least one biomarker.
Measure: Mean (Standard Deviation); unit: Fluorescent Intensity Unit (FIU)
Arm/Group | Active Titration Arm | Placebo Titration Arm | Non-randomized Arm
Number analyzed (Participants) | 17 | 22 | 20
Fluorescent Intensity Unit (FIU)
  Baseline CECs Count (n=17,22,20) | 23584 (18213.1) | 28544 (27694.4) | 29663 (30651.0)
  Baseline MFI PDGFR-BETA (n=17,22,20) | 346815 (179563) | 455238 (238157) | 327567 (167728)
  Baseline MFI pPDGFR-BETA (n=17,22,20) | 401226 (195445) | 395509 (136933) | 397672 (193172)
  Baseline MFI pVEGFR (n=16,22,20) | 456086 (290174) | 436197 (128225) | 398754 (188137)
  Baseline MFI VEGFR (n=16,22,20) | 367799 (181320) | 473290 (228619) | 359092 (167706)

15. Secondary Outcome: Comparison of the Ratio of CECs in Blood: CD146+/CD105+ at Each Time Point to Baseline
Description: CECs are noninvasive marker of vascular damage, remodeling, and dysfunction. Samples were collected and following proteins were analyzed: CD146+/CD105+ CECs, CD146+/CD105+ MFI platelet derived growth factor receptor (PDGFR)-beta, CD146+/CD105+ MFI phospho-PDGFR (pPDGFR)-beta, CD146+/CD105+ phospho-VEGFR (pVEGFR), CD146+/CD105+ MFI VEGFR. The ratio of plasma levels of the biomarkers at the selected time point vs baseline is reported.
Time Frame: At end of the lead-in period (Cycle 1 Day 15), Cycle 2 Day 15 and End of therapy (EOT)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Active Titration Arm | Placebo Titration Arm | Non-randomized Arm
Number analyzed (Participants) | 17 | 22 | 20
Ratio
  C1D15:C1D1 CECs Count (n=11,18,14) | 2.3 (2.52) | 3.7 (6.92) | 2.2 (3.10)
  C2D15:C1D1 CECs Count (n=13,16,11) | 1.3 (1.43) | 4.4 (9.27) | 1.3 (1.22)
  EOT:C1D1 CECs Count (n=7,9,4) | 2.8 (4.81) | 8.9 (21.70) | 1.2 (1.50)
  C1D15:C1D1 MFI PDGFRBETA (n=11,17,13) | 1.3 (1.03) | 1.5 (1.14) | 1.1 (0.73)
  C2D15:C1D1 MFI PDGFRBETA (n=13,16,11) | 1.4 (1.24) | 1.1 (1.14) | 2.2 (1.62)
  EOT:C1D1 MFI PDGFRBETA (n=7,9,4) | 1.5 (1.75) | 0.6 (0.52) | 1.2 (1.78)
  C1D15:C1D1 MFI pPDGFR-BETA (n=11,17,13) | 1.1 (0.63) | 1.2 (0.77) | 1.0 (1.12)
  C2D15:C1D1 MFI pPDGFR-BETA (n=13,16,11) | 1.0 (0.69) | 0.8 (0.45) | 1.2 (0.79)
  EOT:C1D1 MFI pPDGFRBETA (n=7,9,4) | 0.8 (0.71) | 0.8 (0.93) | 1.9 (1.57)
  C1D15:C1D1 MFI pVEGFR (n=10,18,14) | 1.0 (0.46) | 1.2 (0.88) | 1.2 (1.00)
  C2D15:C1D1 MFI pVEGFR (n=12,16,11) | 1.0 (0.74) | 0.9 (0.82) | 1.2 (0.80)
  EOT:C1D1 MFI pVEGFR (n=7,9,4) | 0.8 (0.53) | 1.3 (0.96) | 3.0 (1.16)
  C1D15:C1D1 MFI VEGFR (n=10,18,14) | 1.4 (1.25) | 1.3 (0.94) | 1.0 (0.64)
  C2D15:C1D1 MFI VEGFR (n=12,16,11) | 1.5 (1.48) | 1.3 (0.99) | 2.1 (1.72)
  EOT:C1D1 MFI VEGFR (n=7,9,4) | 1.1 (1.03) | 0.7 (0.48) | 1.9 (1.63)

16. Secondary Outcome: Circulating Endothelial Cells (CECs) in Blood: CD31+/CD146+
Description: CECs are noninvasive marker of vascular damage, remodeling, and dysfunction. Samples were collected and following proteins were analyzed: CD31+/CD146+ CECs, CD31+/CD146+ MFI PDGFR-beta, CD31+/CD146+ MFI pPDGFR-beta, CD31+/CD146+ pVEGFR, CD31+/CD146+ MFI VEGFR. The ratio of plasma levels of the biomarkers at the selected time point vs baseline is reported.
Time Frame: At baseline - Beginning of the lead-in period (Cycle 1 Day 1)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Fluorescent Intensity Unit (FIU)
Arm/Group | Active Titration Arm | Placebo Titration Arm | Non-randomized Arm
Number analyzed (Participants) | 17 | 22 | 20
Fluorescent Intensity Unit (FIU)
  Baseline CECs Count (n=17,22,20) | 74668 (50558.9) | 76258 (46779.5) | 77437 (63419.4)
  Baseline MFI PDGFR-BETA (n=17,21,20) | 333760 (164604) | 380886 (147261) | 442642 (267436)
  Baseline MFI pPDGFR-BETA (n=17,21,20) | 380139 (205600) | 355441 (147046) | 383202 (211174)
  Baseline MFI pVEGFR (n=17,22,20) | 385617 (203956) | 352644 (128803) | 380184 (173578)
  Baseline MFI VEGFR (n=17,22,20) | 330333 (151710) | 401909 (165235) | 359097 (146943)

17. Secondary Outcome: Comparison of Ratio of CECs in Blood: CD31+/CD146+ at Each Time Point to Baseline
Description: as for outcome 16
Time Frame: At end of the lead-in period (Cycle 1 Day 15), Cycle 2 Day 15 and End of therapy (EOT)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Active Titration Arm | Placebo Titration Arm | Non-randomized Arm
Number analyzed (Participants) | 17 | 22 | 20
Ratio
  C1D15:C1D1 CECs Count (n=11,18,14) | 2.7 (3.17) | 1.6 (2.32) | 1.5 (2.31)
  C2D15:C1D1 CECs Count (n=13,16,11) | 1.4 (1.38) | 2.2 (3.91) | 2.5 (3.98)
  EOT:C1D1 CECs COUNT (n=7,9,4) | 1.5 (1.95) | 1.4 (2.66) | 0.6 (0.71)
  C1D15:C1D1 MFI PDGFRBETA (n=11,15,13) | 1.2 (0.74) | 1.3 (0.89) | 0.8 (0.51)
  C2D15:C1D1 MFI PDGFRBETA (n=13,14,11) | 1.4 (1.36) | 1.1 (1.03) | 2.2 (2.64)
  EOT:C1D1 MFI PDGFRBETA (n=6,8,4) | 1.2 (1.23) | 0.6 (0.51) | 1.7 (1.49)
  C1D15:C1D1 MFI pPDGFR-BETA (n=11,15,13) | 1.2 (1.07) | 1.4 (0.81) | 1.0 (0.87)
  C2D15:C1D1 MFI pPDGFR-BETA (n=13,14,11) | 1.2 (0.89) | 0.8 (0.38) | 1.1 (0.71)
  EOT:C1D1 MFI pPDGFRBETA (n=6,8,4) | 0.7 (0.63) | 0.8 (0.91) | 3.0 (0.47)
  C1D15:C1D1 MFI pVEGFR (n=11,18,14) | 1.1 (0.75) | 1.4 (0.74) | 1.2 (0.90)
  C2D15:C1D1 MFI pVEGFR (n=13,16,10) | 1.2 (1.00) | 0.9 (0.68) | 1.3 (0.70)
  EOT:C1D1 MFI pVEGFR (n=7,9,4) | 0.7 (0.59) | 1.1 (1.24) | 3.1 (0.95)
  C1D15:C1D1 MFI VEGFR (n=11,18,14) | 1.3 (0.93) | 1.3 (0.90) | 1.0 (0.57)
  C2D15:C1D1 MFI VEGFR n=13,16,10) | 1.5 (1.44) | 1.2 (0.96) | 2.1 (1.80)
  EOT:C1D1 MFI VEGFR (n=7,9,4) | 1.2 (1.27) | 1.1 (0.90) | 1.5 (1.42)

18. Secondary Outcome: ORR in Subgroups That Were Defined by Vascular Endothelial Growth Factor A (VEGFA) or Vascular Endothelial Growth Factor Receptor 3 (VEGFR3) Polymorphisms
Description: ORR, defined as proportion of participants with CR or PR according to RECIST, in subgroups that were defined by VEGFA or VEGFR3 polymorphisms.
Time Frame: At baseline - Beginning of the lead-in period (Cycle 1 Day 1)
Population: The Safety Analysis (SA) population consisted of all participants who received at least one dose of study medication with treatment assignments designated according to actual study treatment received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Active Titration Arm | Placebo Titration Arm | Non-randomized Arm
Number analyzed (Participants) | 49 | 49 | 79
Percentage of participants
  VEGFA/rs699947 Genotype: A/A (n = 7, 9, 14) | 85.7 [42.1 to 99.6] | 22.2 [2.8 to 60.0] | 42.9 [17.7 to 71.1]
  VEGFA/rs699947 Genotype: A/C (n = 22, 20, 41) | 54.5 [32.2 to 75.6] | 35.0 [15.4 to 59.2] | 65.9 [49.4 to 79.9]
  VEGFA/rs699947 Genotype: C/C (n = 14, 14, 24) | 50.0 [23.0 to 77.0] | 35.7 [12.8 to 64.9] | 66.7 [44.7 to 84.4]
  VEGFA/rs1570360 Genotype: G/G (n = 22, 23, 43) | 59.1 [36.4 to 79.3] | 39.1 [19.7 to 61.5] | 67.4 [51.5 to 80.9]
  VEGFA/rs1570360 Genotype: G/A (n = 19, 16, 29) | 57.9 [33.5 to 79.7] | 18.8 [4.0 to 45.6] | 58.6 [38.9 to 76.5]
  VEGFA/rs1570360 Genotype: A/A (n = 2, 4, 7) | 50.0 [1.3 to 98.7] | 50.0 [6.8 to 93.2] | 42.9 [9.9 to 81.6]
  VEGFR3/rs448012 Genotype: G/G (n = 16, 15, 28) | 81.3 [54.4 to 96.0] | 53.3 [26.6 to 78.7] | 60.7 [40.6 to 78.5]
  VEGFR3/rs448012 Genotype: G/C (n = 22, 22, 35) | 45.5 [24.4 to 67.8] | 18.2 [5.2 to 40.3] | 57.1 [39.4 to 73.7]
  VEGFR3/rs448012 Genotype: C/C (n = 5, 6, 16) | 40.0 [5.3 to 85.3] | 33.3 [4.3 to 77.7] | 75.0 [47.6 to 92.7]
  VEGFR3/rs307826 Genotype: A/A (n = 36, 39, 79) | 58.3 [40.8 to 74.5] | 30.8 [17.0 to 47.6] | 64.3 [51.9 to 75.4]
  VEGFR3/rs307826 Genotype: A/G (n = 6, 4, 9) | 50.0 [11.8 to 88.2] | 50.0 [6.8 to 93.2] | 44.4 [13.7 to 78.8]
  VEGFR3/rs307826 Genotype: G/G (n = 1, 0, 0) | 100.0 [2.5 to 100.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  VEGFR3/rs307821 Genotype: G/G (n = 36, 38, 79) | 55.6 [38.1 to 72.1] | 28.9 [15.4 to 45.9] | 65.2 [52.8 to 76.3]
  VEGFR3/rs307821 Genotype: G/T (n = 6, 5, 10) | 66.7 [22.3 to 95.7] | 60.0 [14.7 to 94.7] | 40.0 [12.2 to 73.8]
  VEGFR3/rs307821 Genotype: T/T (n = 1, 0, 0) | 100.0 [2.5 to 100.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]

19. Secondary Outcome: PFS in Subgroups That Were Defined by Vascular Endothelial Growth Factor A (VEGFA) or Vascular Endothelial Growth Factor Receptor 3 (VEGFR3) Polymorphisms
Description: PFS, defined as the time from randomization to first documentation of objective tumor progression or to death due to any cause, in subgroups that were defined by VEGFA or VEGFR3 polymorphisms. Estimates of the PFS curves from the Kaplan-Meier method were presented.
Time Frame: At baseline - Beginning of the lead-in period (Cycle 1 Day 1)
Population: as for outcome 18
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Active Titration Arm | Placebo Titration Arm | Non-randomized Arm
Number analyzed (Participants) | 43 | 43 | 79
Months
  VEGFA/rs699947 Genotype: A/A (n = 7, 9, 14) | NA [1.74 to NA] — Values were not calculable due to the large number of censored event times | 11.50 [3.58 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times | 7.33 [5.06 to 13.83]
  VEGFA/rs699947 Genotype: A/C (n = 22, 20, 41) | 11.07 [3.02 to 17.44] | 9.67 [1.91 to 16.59] | 16.59 [10.97 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times
  VEGFA/rs699947 Genotype: C/C (n = 14, 14, 41) | 18.74 [1.84 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times | 24.64 [4.01 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times | 25.13 [8.28 to 30.45]
  VEGFA/rs1570360 Genotype: G/G (n = 22, 23, 43) | 14.62 [7.39 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times | 19.42 [5.81 to 27.63] | 25.13 [11.47 to 30.45]
  VEGFA/rs1570360 Genotype: G/A (n = 19, 16, 29) | 12.78 [1.84 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times | 8.34 [1.91 to 16.59] | 13.90 [8.28 to 22.54]
  VEGFA/rs1570360 Genotype: A/A (n = 2, 4, 29) | NA [1.74 to NA] — Values were not calculable due to the large number of censored event times | 10.04 [3.58 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times | 8.57 [1.74 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times
  VEGFR3/rs448012 Genotype: G/G (n = 16, 15, 28) | 17.44 [12.78 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times | 19.42 [5.35 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times | 22.54 [8.08 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times
  VEGFR3/rs448012 Genotype: G/C (n = 22, 22, 35) | 9.18 [1.84 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times | 8.31 [3.58 to 16.52] | 13.83 [5.62 to 16.59]
  VEGFR3/rs448012 Genotype: C/C (n = 5, 6, 16) | 11.07 [1.84 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times | 15.67 [1.91 to 27.63] | NA [8.57 to NA] — Values were not calculable due to the large number of censored event times
  VEGFR3/rs307826 Genotype: A/A (n = 36, 39, 70) | 13.73 [8.28 to 24.47] | 15.67 [8.21 to 22.17] | 16.56 [10.28 to 25.13]
  VEGFR3/rs307826 Genotype: A/G (n = 6, 4, 9) | 16.52 [1.18 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times | 7.93 [1.84 to 11.86] | 16.26 [2.66 to 30.45]
  VEGFR3/rs307826 Genotype: G/G (n = 0, 0, 0) | NA [NA to NA] — Number of participants with an event in this category was 0 | NA [NA to NA] — Number of participants with an event in this category was 0 | NA [NA to NA] — Number of participants with an event in this category was 0
  VEGFR3/rs307821 Genotype: G/G (n = 36, 38, 69) | 12.78 [7.39 to 24.47] | 15.67 [8.21 to 23.95] | 16.59 [10.28 to 28.52]
  VEGFR3/rs307821 Genotype: G/T (n = 36, 38, 10) | 24.80 [1.18 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times | 8.34 [1.84 to 11.86] | 13.86 [2.66 to 30.45]
  VEGFR3/rs307821 Genotype: T/T (n = 1, 0, 0) | NA [NA to NA] — Number of participants with an event in this category was 1 | NA [NA to NA] — Number of participants with an event in this category was 0 | NA [NA to NA] — Number of participants with an event in this category was 0

ADVERSE EVENTS:
Time Frame: AEs were reported until follow up visit. Non-SAEs: up to 28 days post last dose or upon starting new anticancer treatment, whichever was first. SAEs: up to 28 days post last dose, irrespective of new anticancer treatment.
Description: The same event may be referred to as (serious and non-serious) AEs. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Discontinued Prior to Randomization: Participants who were discontinued prior to randomization to either treatment or non-randomization arms.
Arm/Group | Active Titration Arm | Placebo Titration Arm | Non-randomized Arm | Discontinued Prior to Randomization
Serious Adverse Events (participants affected / at risk) | 25/56 | 14/56 | 39/91 | 2/10
Other Adverse Events (participants affected / at risk) | 55/56 | 51/56 | 91/91 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Active Titration Arm (N=56) | Placebo Titration Arm (N=56) | Non-randomized Arm (N=91) | Discontinued Prior to Randomization (N=10)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 2 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 4 | 0 | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 0 | 1 | 0/1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Disease progression (General disorders) | 1 | 1 | 6 | 0
General physical health deterioration (General disorders) | 1 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 1 | 0 | 0
Lung abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 2 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 0 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Postrenal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 2 | 0
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Incisional hernia repair (Surgical and medical procedures) | 0 | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Monoparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Titration Arm (N=56) | Placebo Titration Arm (N=56) | Non-randomized Arm (N=91) | Discontinued Prior to Randomization (N=10)
Anaemia (Blood and lymphatic system disorders) | 5 | 4 | 9 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 2
Hypothyroidism (Endocrine disorders) | 18 | 13 | 41 | 2
Abdominal pain (Gastrointestinal disorders) | 9 | 9 | 11 | 1
Abdominal pain upper (Gastrointestinal disorders) | 6 | 2 | 11 | 0
Constipation (Gastrointestinal disorders) | 11 | 7 | 27 | 3
Diarrhoea (Gastrointestinal disorders) | 34 | 35 | 58 | 1
Dry Mouth (Gastrointestinal disorders) | 7 | 2 | 7 | 0
Dyspepsia (Gastrointestinal disorders) | 7 | 5 | 18 | 0
Flatulence (Gastrointestinal disorders) | 7 | 3 | 4 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 1 | 4 | 1
Nausea (Gastrointestinal disorders) | 24 | 19 | 33 | 2
Stomatitis (Gastrointestinal disorders) | 10 | 4 | 17 | 0
Vomiting (Gastrointestinal disorders) | 18 | 12 | 25 | 2
Asthenia (General disorders) | 6 | 5 | 6 | 0
Fatigue (General disorders) | 27 | 26 | 49 | 4
Mucosal inflammation (General disorders) | 12 | 8 | 13 | 0
Rhinitis (Infections and infestations) | 3 | 6 | 4 | 0
Alanine aminotransferase increased (Investigations) | 6 | 9 | 12 | 0
Aspartate aminotransferase increased (Investigations) | 6 | 10 | 12 | 0
Blood creatinine increased (Investigations) | 4 | 8 | 14 | 1
Blood glucose increased (Investigations) | 4 | 7 | 10 | 2
Fibrin D dimer increased (Investigations) | 0 | 1 | 0 | 1
Weight decreased (Investigations) | 16 | 12 | 25 | 1
Decreased appetite (Metabolism and nutrition disorders) | 21 | 16 | 37 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 11 | 17 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 8 | 17 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 4 | 15 | 0
Dysgeusia (Nervous system disorders) | 9 | 5 | 21 | 1
Headache (Nervous system disorders) | 9 | 15 | 27 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 4 | 1
Paraesthesia (Nervous system disorders) | 5 | 3 | 3 | 1
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 3 | 4 | 8 | 1
Haemoglobinuria (Renal and urinary disorders) | 2 | 3 | 5 | 1
Proteinuria (Renal and urinary disorders) | 12 | 12 | 40 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 19 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 18 | 20 | 44 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 8 | 27 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 3 | 7 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 18 | 10 | 40 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 6 | 13 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 8 | 19 | 0
Hypertension (Vascular disorders) | 35 | 24 | 76 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 3 | 15 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 3 | 3 | 0
Gastritis (Gastrointestinal disorders) | 3 | 2 | 9 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3 | 6 | 0
Oedema peripheral (General disorders) | 4 | 3 | 14 | 0
Pain (General disorders) | 4 | 3 | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 6 | 0
Blood alkaline phosphatase increased (Investigations) | 4 | 4 | 6 | 2
Blood glucose decreased (Investigations) | 3 | 5 | 1 | 0
Blood potassium increased (Investigations) | 4 | 3 | 4 | 0
Blood thyroid stimulating hormone increased (Investigations) | 8 | 7 | 9 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 1 | 5 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 7 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 9 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 4 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 8 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 9 | 23 | 2
Dizziness (Nervous system disorders) | 8 | 10 | 14 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 12 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 8 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 3 | 14 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 3 | 4 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 6 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 2 | 1
Proctalgia (Gastrointestinal disorders) | 2 | 0 | 5 | 0
Toothache (Gastrointestinal disorders) | 1 | 3 | 5 | 0
Chest pain (General disorders) | 5 | 2 | 6 | 0
Chills (General disorders) | 4 | 1 | 5 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 6 | 3 | 4 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 1 | 5 | 0
Nasopharyngitis (Infections and infestations) | 4 | 3 | 19 | 0
Respiratory tract infection (Infections and infestations) | 2 | 3 | 0 | 0
Sinusitis (Infections and infestations) | 4 | 2 | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 10 | 1
Blood albumin decreased (Investigations) | 1 | 3 | 1 | 0
Blood sodium decreased (Investigations) | 2 | 3 | 1 | 0
Blood triglycerides increased (Investigations) | 2 | 2 | 5 | 0
Haemoglobin decreased (Investigations) | 1 | 1 | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 4 | 5 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 3 | 6 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 3 | 6 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 1 | 3 | 0
Anxiety (Psychiatric disorders) | 3 | 3 | 7 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 4 | 4 | 6 | 0
Dysuria (Renal and urinary disorders) | 3 | 0 | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 6 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 4 | 5 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 3 | 1 | 0
Hypotension (Vascular disorders) | 0 | 8 | 9 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.